CLINICAL TRIAL: NCT05560087
Title: Association of PeRiODontal Disease and gUt Microbiome With Coronary artEry Disease (PRODUCE Study)
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0533
Record Dates: First submitted 2022-09-19; First posted 2022-09-29 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis; Coronary Heart Disease; Human Microbiome; Dysbiosis
MeSH Terms: conditions — Periodontitis; Coronary Disease; Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Stool, and Gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary artery disease
- control

SUMMARY:
The purpose of this study is to explore the relationship between periodontal disease and coronary artery disease through changes in the gut microbiome. In addition, the investigators aim to find possible periodontal pathogens that have association with cardiovascular disease.

DETAILED DESCRIPTION:
The previous studies have reported the associations among cardiovascular disease, periodontitis, and gut microbiome dysbiosis. However, there is a lack of evidences about the axis of association from oral-gut-cardiovascular disease. The investigators hypothesized that periodontal disease might induce dysbiosis of gut microbiome and dysbiosis might have a role in cardiovascular disease (as called "oro-gut-vascular axis"). The investigators aim to prove this hypothesis through this case-control, cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

-Patients aged from 19 to 80 years who underwent invasive coronary angiography for clinical necessity, with informed consent

Exclusion Criteria:

* Patients with prosthetic valve
* pregnancy
* active malignancy
* active autoimmune disease
* active inflammatory bowel disease
* chronic kidney disease (eGFR<30, or on dialysis)
* Active liver disease or liver cirrhosis
* consistent use of probiotics
* prior gastrointestinal surgery within 1 year

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged from 19 to 80 years who underwent invasive coronary angiography for clinical necessity in single tertiary hospital
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
The association between periodontal disease and cardiovascular disease | within 3 years after enrollment (until the completion of dataset)
  The association between periodontal disease and cardiovascular disease by chi-square test The difference of relative abundance in gut microbiome by PERMANOVA test Safety Issue: No

SECONDARY OUTCOMES:
The associations among periodontitis, gut microbiome and biomarkers | within 3 years after enrollment (until the completion of dataset)
  The association between periodontal disease and biomarkers by independent t-test
The associations between periodontitis and cognitive function | within 3 years after enrollment (until the completion of dataset)
  The associtation between periodontal disease and cognitive function by chi-square test

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Won Ha, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea